CLINICAL TRIAL: NCT05711173
Title: Role of Clonal Hematopoiesis and NETs Formation in Unusual Venous Thrombosis (CLODETTE)
Brief Title: Clonal Hematopoiesis and NETs Formation in Venous Thrombosis (CLODETTE)
Acronym: CLODETTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2022/32
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Venous Thromboses; Thromboembolic Disease; Neutrophil Extracellular Trap Formation; Clonal Hematopoiesis of Indeterminate Potential
Keywords: Thrombosis; Venous thrombosis; Clonal hematopoiesis of indetermined potential
MeSH Terms: conditions — Venous Thrombosis; Thromboembolism; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Additional blood sampling — The procedure will consist of an additional blood sample for ETDA tube collection (NGS analysis) and citrate tube collection (NETose analysis)

SUMMARY:
Thrombo-embolic venous diseases are represented by deep venous thrombosis and/or pulmonary embolism. In some patients with repeated thrombosis or occurrence of thrombosis in unusual sites, the etiological workup remains negative, which represents a problem for the management of the anticoagulant treatments. Recently, two factors have been identified as important in the physiopathology of hemostasis and coagulation: the presence of clonal hematopoiesis of indetermined potential (CHIP) and the formation of neutrophil extracellular traps (NETs). In this study, these two factors will be studied in patients with repeated venous thrombosis or thrombosis occurring in unusual site.

DETAILED DESCRIPTION:
It has recently been shown that some patients clonal have mutations at a low level in hematopoietic cells (this phenomenon is named clonal hematopoiesis of indetermined potential (CHIP)) and that the presence of a clonal hematopoiesis is associated with an increased cardiovascular risk. However, few data exist about the implication of CHIP in venous thrombosis. Neutrophils extracellular traps are involved in the activation of hemostasis and coagulation. Murine models have highlighted the crucial role of NETs in the physiopathology of venous thrombosis. In patients, studies have demonstrated that NETs markers were present in arteries lesions as coronary plaques. However, few studies have analyzed the NETosis in the setting of venous thrombosis.

The study hypothesis is that patients with venous thrombosis may have an increased prevalence of CHIP and/or an increased NETosis formation, which may represent a predisposition for the occurrence of venous thrombosis. We also speculate that patients with CHIP may have an increased NETosis, due to the presence of activating clonal mutations in neutrophils.

Patients included will be : younger than 50-years-old with repeated thrombosis or thrombosis of unusual sites (cerebral venous thrombosis, splanchnic thrombosis) with a negative etiological workup and notably the absence of constitutional or acquired venous thrombosis risk factors. In this population, we will analyze the prevalence of CHIP and the NETosis via the study of 4 different NETosis plasmatic markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) less than 50 y.o with :
* Splanchnic venous territory thrombosis or
* Cerebral venous thrombosis or
* Venous thrombosis of the upper limb or
* Pulmonary embolism (1st episode if male, 2nd episode if female) unprovoked or
* 1 episode of deep vein thrombosis + 1 episode of arterial thrombosis

Exclusion Criteria:

* Presence of a major or minor transient venous thrombosis risk factor:
* Surgery within the last 3 months preceding the qualifying thrombotic episode
* Lower limb fracture with immobilization > 3 days in the last 3 months preceding the qualifying thrombotic episode
* Presence of estro-progestational contraception
* Pregnancy
* Immobilization for acute medical reasons within the last 3 months preceding the qualifying thrombotic episode
* Air or car travel > 6 hours
* Presence of a major or minor persistent risk factor for venous thrombosis:
* Presence of active cancer (solid cancer or hematologic malignancy)
* Chronic inflammatory digestive or joint diseases
* Ongoing treatment with heparin (low molecular weight heparin (LMWH) or unfractionated heparin (UFH))
* Presence of an abnormality on the thrombophilia test among the following abnormalities
* Protein C deficiency
* Protein S deficiency
* Anti-thrombin deficiency
* Heterozygous or homozygous factor II mutation
* Heterozygous or homozygous factor V mutation
* Presence of anti-phospholipid syndrome
* Presence of myeloproliferative neoplasia
* Presence of paroxysmal nocturnal hemoglobinuria

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Presence of clonal hematopoiesis | At baseline
  The existence of clonal hematopoiesis will be defined as the demonstration of at least one mutation in the blood cells of an apparently healthy subject (without obvious hematological pathology). DNA will be extracted from circulating leukocytes to search for mutations in a panel of 59 genes

SECONDARY OUTCOMES:
Presence of one or more increased NETosis markers and/or a decreased NETosis-inhibiting marker (DNAse level) compared to a control population. | At baseline
  Analysis of the following markers: MPO-DNA complex, Histone 3-DNA complex, citrullinated histone 3, DNAse
Correlation (correlation coefficient values) between the presence of a CHIP and the formation of NETs | During final analysis
  Correlation analysis will be performed between each NETosis marker and CHIP evaluation (presence or absence, number of mutations, variant allele frequency for each mutation)
Allele frequency | At baseline
  Variant allele frequency of each detected mutation will be determined using NGS analysis
Number of clonal mutations | At baseline
  The number of clonal mutations for each patient will be determined using NGS analysis
C-reactive protein (CRP) level as a marker of inflammation | At baseline
  C-reactive protein concentration will be determined for each patient, as a marker of inflammation
Site(s) of thrombosis | At baseline
  Site(s) of thrombosis will be determined during examination of the patient
Number of thrombosis | At baseline
  The number of thrombosis will be determined during examination of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre GUY, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - CHU de Bordeaux, Service de Neurologie, Bordeaux
  - CHU de Bordeaux, Service Gastro-Entérologie, Bordeaux
  - CHU de Bordeaux, Service Hématologie Biologique, Bordeaux
  - CHU de Bordeaux, Service Médecine Vasculaire, Bordeaux
  - CHU de Bordeaux, Unité ambulatoire de Médecine Vasculaire, Bordeaux
  - CHU de Lille, Service Hémostase Clinique, Lille
  - APHM - Hôpital de la Timone, Service Hématologie, Marseille